CLINICAL TRIAL: NCT06000358
Title: The Effect of Combined Cryotherapy and Immunotherapy on Systemic T Cell Changes and Clinical Outcomes in Metastatic Non-small Cell Lung Cancer
Acronym: LUCACRIMUNO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Research Council of Lithuania (Other)
Responsible Party: Principal Investigator, Marius Zemaitis, Professor, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUCACRIMUNO-001
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer Stage IV
Keywords: Pulmonology; Oncology; Immunotherapy; Cryotherapy
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — pembrolizumab; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cryotherapy and Pembrolizumab monotherapy; (Active Comparator): Patients with metastatic non-small cell lung cancer, who are eligible for first-line pembrolizumab monotherapy (PD-L1 expression equal to or greater than 50%, no EGFR mutations or ALK translocations). Bronchoscopic cryotherapy procedure is performed before the start of systemic treatment.
  Interventions: Procedure: Bronchoscopic cryotherapy; Drug: Pembrolizumab
- Cryotherapy and Pembrolizumab with platinum-based chemotherapy; (Active Comparator): Patients with metastatic non-small cell lung cancer, who are eligible for first-line pembrolizumab and platinum-based chemotherapy (PD-L1 expression less than 50%, no EGFR mutations or ALK translocations). Bronchoscopic cryotherapy procedure is performed before the start of systemic treatment.
  Interventions: Procedure: Bronchoscopic cryotherapy; Drug: Pembrolizumab; Drug: Platinum based chemotherapy
- Pembrolizumab monotherapy; (Active Comparator): Patients with metastatic non-small cell lung cancer, who are eligible for first-line pembrolizumab monotherapy (PD-L1 expression equal to or greater than 50%, no EGFR mutations or ALK translocations).
  Interventions: Drug: Pembrolizumab
- Pembrolizumab with platinum-based chemotherapy; (Active Comparator): Patients with metastatic non-small cell lung cancer, who are eligible for first-line pembrolizumab and platinum-based chemotherapy (PD-L1 expression less than 50%, no EGFR mutations or ALK translocations).
  Interventions: Drug: Pembrolizumab; Drug: Platinum based chemotherapy

INTERVENTIONS:
Procedure: Bronchoscopic cryotherapy — The cryotherapy procedure is performed before the start of systemic treatment, under visual (for endobronchial cryotherapy) or radial EBUS and fluoroscopy control (for transbronchial cryotherapy), ensuring the correct position of the cryoprobe in the tumor. After being placed in the correct position. After being placed in the correct position, the cryoprobe is cooled using CO2 and allowed to cool passively. The cooling-thawing stages are repeated for a total of 3 cycles.
  Arms: Cryotherapy and Pembrolizumab monotherapy;; Cryotherapy and Pembrolizumab with platinum-based chemotherapy;
Drug: Pembrolizumab — As a standard of care, patients will receive pembrolizumab.
Drug: Platinum based chemotherapy — As a standard of care, patients will receive platinum-based chemotherapy in addition to pembrolizumab if PD-L1 expression is less than 50%.
  Arms: Cryotherapy and Pembrolizumab with platinum-based chemotherapy;; Pembrolizumab with platinum-based chemotherapy;

SUMMARY:
Lung cancer remains one of the most commonly diagnosed oncological diseases worldwide and the first in terms of mortality. Although immune checkpoint inhibitors form the backbone of current metastatic non-small cell lung cancer treatments, there is still no ideal predictive marker for its efficacy and patients still achieve suboptimal results in overall response and survival. While immune checkpoint inhibitors are known to shift systemic anti-tumor immune response from suppression to stimulation in some patients, the investigators hypothesize that this effect can be further enhanced by cryotherapy, especially in "cold" tumors. If proven successful, cryotherapy in combination with immunotherapy, could potentiate a more powerful immune response compared to systemic therapy alone, improve overall response rate, patients' survival without disease progression, and overall survival. The investigators, therefore, aim to use combined local tumor cryotherapy, combined with immune checkpoint inhibitor therapy to induce and evaluate systemic anti-tumor T lymphocyte response and achieve improved non-small cell lung cancer patient outcomes than with immunotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Eastern Cooperative Oncology Group (ECOG) performance score 0 - 1;
* Patients with histologically confirmed metastatic non-small cell lung cancer and PD-L1 expression on tumor cells was evaluated;
* CT examination shows measurable tumor formations according to the RECIST 1.1 criteria;
* Primary lung tumor or metastasis accessible to flexible bronchoscopy;
* Patients may have received surgery, adjuvant or neoadjuvant chemotherapy prior to the study if it was completed at least 12 months before relapse;
* Patients informed about the purpose and course of the study and provided a written consent to participate.

Exclusion Criteria:

* Patients who refused to participate in the clinical trial and did not sign the informed consent form;
* Men and women under the age of 18, pregnant women;
* Patients belonging to a vulnerable social group;
* High risk of general anesthesia, defined as American Society of Anesthesiologists (ASA) class 4 - 6;
* Documented allergy to medications used during general and local anesthesia, systemic cancer treatment;
* Patients previously treated with immune checkpoint inhibitors;
* EGFR mutations or ALK translocations have been identified in patients;
* Patients with previously diagnosed autoimmune diseases, active viral hepatitis, uncontrolled human immunodeficiency virus (HIV) infection or untreated tuberculosis;
* Patients treated with immunosuppressive drugs, systemic corticosteroids, with equivalent doses of prednisolone exceeding 10 mg/day;
* Patients with an increased risk of bleeding during an interventional procedure;
* Acute untreated conditions that would make it impossible to perform an interventional lung procedure.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in T Lymphocyte Count and Function in Response to Cryotherapy and Immunotherapy | 6 weeks
  Changes in T lymphocyte counts and function in peripheral venous blood assessed via flow cytometry

SECONDARY OUTCOMES:
Necrotic cancer cell death | 6 weeks
  A change in the concentration of High mobility group box 1 protein (HMGB-1) in venous blood
The influence of immune cell infiltration in tumor tissue on subsequent cryotherapy and immunotherapy treatment | 1 day
  Number of tumor-infiltrating CD4 and CD8 lymphocytes in non-small cell lung cancer biopsy material by immunohistochemistry.
Objective response rate | 1 year
  Assessed according to RECIST and iRECIST criteria
Progression-free survival | 1 year
  The time from the first cycle of systemic treatment to radiologically confirmed disease progression
Overall survival | 1 year
  The time from the first cycle of systemic treatment to death from any cause
Safety of bronchoscopic cryotherapy and immunotherapy | 1 year
  Documentation and assessment of adverse treatment events according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Changes in T Lymphocyte Function in Response to Cryotherapy and Immunotherapy | 6 weeks
  Changes in T lymphocyte function in peripheral venous blood assessed via RNA expression
Changes in T Lymphocyte Effector Function in Response to Cryotherapy and Immunotherapy | 6 weeks
  Changes in T lymphocyte effector function in peripheral venous blood evaluated via cytokine panels

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania